CLINICAL TRIAL: NCT05995639
Title: Comparison of the Effects of Dry Needling and Ozone Treatment on Pain and Functionality in Myofascial Pain Syndrome of the Upper Trapezius
Brief Title: Dry Needling Versus Ozone in Myofascial Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uskudar State Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Hüseyin Temel, Principal Investigator, Uskudar State Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DnvsO
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Dry Needling; Ozone; Trapezius; Trigger Point Pain, Myofascial; Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Dry Needling; Ozone

STUDY DESIGN:
Intervention Model Description: In this prospective randomized study to be conducted in Üsküdar state hospital, patients diagnosed with myofascial pain syndrome in the upper part of the trapezius muscle will be divided into 3 equal groups.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators and outcomes assessors will be blinded to the procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Patients who will undergo an exercise treatment for the UT. The exercise therapy will focus on stretching exercises for the UT. Exercise therapy will undergo 2 weeks.
- Dry Needling Group (Active Comparator): Patients who will undergo DN treatment for the UT. A clinician with 5 years of DN experience will assess patients and apply DN treatment. The active trigger points will be diagnosed by the criteria described by Simons and Travell. 0.25x25mm acupuncture needles will be used. DN will be performed with fast in fast out technique and needling will continue until a local twitch response is elicited. Treatment will be applied 3 times, one week apart.
  Interventions: Procedure: Dry Needling
- Ozone Group (Active Comparator): Patients who will undergo ozone treatment for the UT. A clinician with 10 years of ozone experience will assess patients and apply ozone treatment. 12 gamma ozone will be used. Patients will be injected with ozone in UT with most sensitive parts. Treatment will be applied 3 times, one week apart.
  Interventions: Procedure: Ozone Injection

INTERVENTIONS:
Procedure: Dry Needling — Dry needling is an evidence-based therapeutic procedure used primarily in musculoskeletal rehabilitation. It involves inserting thin needles into specific trigger points in muscles, tendons, or fascia, aiming to alleviate pain and improve musculoskeletal function. Unlike acupuncture, dry needling focuses on resolving myofascial pain and dysfunction by directly targeting trigger points, often identified through palpation and anatomical understanding. Academic exploration of dry needling delves into its physiological mechanisms, clinical effectiveness, and potential integration into comprehensive treatment strategies.
  Arms: Dry Needling Group
Procedure: Ozone Injection — Intramuscular ozone injection is a therapeutic intervention utilized within the context of musculoskeletal care, particularly for individuals grappling with conditions such as myofascial pain syndrome and related neuromuscular issues. This technique involves the controlled introduction of ozone gas, a chemically reactive form of oxygen, directly into targeted muscle tissue through an injection. This intramuscular administration is guided by precise anatomical knowledge and is designed to harness the potential therapeutic benefits of ozone's reactive properties.
  Arms: Ozone Group

SUMMARY:
The aim of this study is to compare the effects of dry needling treatment (DN) and ozone treatment on pain and functionality in individuals with myofascial pain syndrome affecting the upper trapezius (UT) region.

DETAILED DESCRIPTION:
In this prospective randomized study to be conducted in Üsküdar state hospital, patients diagnosed with myofascial pain syndrome in the upper part of the trapezius muscle will be divided into 3 groups. 1st group patients will be given stretching exercises for the upper part of the trapezius muscle. The exercise program will last 15 days. In addition to exercise therapy, the 2nd group will receive dry needling treatment using acupuncture needles of 0.25 x 25mm in size by a physical medicine and rehabilitation specialist with 5 years of experience in the field. Active trigger points will be treated. Trigger points will be diagnosed according to the criteria determined by Simons and Travell. Dry needling treatment will be applied in 3 sessions, one week apart. In the 3rd group, in addition to exercise therapy, 10 gamma ozone will be applied in a total of 3 sessions, one week apart to the upper part of the trapezius muscle by a physical therapist with 10 years of experience in the field. Patients will be evaluated at the beginning of the treatment, after 1 week, at the 3rd week, and after 1 month.

ELIGIBILITY:
Inclusion Criteria:

Adults (18-65 years) with diagnosed myofascial pain syndrome affecting the upper trapezius area Willing and able to provide informed consent Able to comprehend and complete study-related assessments Diagnosed with myofascial pain syndrome affecting the upper trapezius area, based on clinical assessment and Simons and Travell criteria No prior exposure to dry needling or ozone therapy for myofascial pain syndrome Medically stable and cleared by a physician for study participation No active musculoskeletal injuries or conditions in the upper trapezius area No participation in similar interventions within the last 6 months

Exclusion Criteria:

Individuals with known contraindications to dry needling or ozone therapy Severe cardiovascular conditions or uncontrolled hypertension Active infections or skin conditions at treatment sites Known bleeding disorders or anticoagulant use Diagnosed with any other chronic pain syndrome not related to myofascial pain syndrome Any ongoing litigation or compensation claims related to pain conditions Recent trauma or surgery in the upper trapezius area Previous adverse reactions to dry needling or ozone therapy Participation in other investigational studies within the last 3 months History of psychological conditions that might interfere with assessment Pregnant or breastfeeding History of malignancy or immunocompromised status Neurological disorders affecting upper trapezius function Severe cognitive impairments that hinder assessment Inability to commit to the study duration or follow-up assessments Any change in medication regimen that might impact pain or functionality during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-02 (Estimated)

PRIMARY OUTCOMES:
Pain measured by Visual Analog Scale | First day, after first week, after three weeks, after one month
  The Visual Analog Scale (VAS) is a widely used pain assessment tool in clinical settings. It involves a simple linear scale typically ranging from 0 to 10, where individuals mark a point to indicate their pain intensity level. The left end of the scale represents "no pain," assigned a value of 0, while the right end corresponds to "worst possible pain," denoted as 10. By gauging pain subjectively through this visual representation, the VAS provides a quantifiable measure of pain intensity, enabling healthcare professionals to track changes in pain over time and tailor treatment strategies accordingly.
Quality of Life Measured by Neck Disability Index | First day, after first week, after three weeks, after one month
  The Neck Disability Index (NDI) is a widely used tool to assess the impact of neck-related conditions on an individual's quality of life. It consists of a questionnaire that comprises ten items, each addressing different aspects of daily functioning and discomfort related to neck pain. Participants rate their level of difficulty in various activities such as lifting, reading, and sleeping on a scale from 0 to 5. The total score is then calculated and expressed as a percentage, providing valuable insights into the extent of neck-related disability and its effect on overall quality of life. The NDI aids clinicians in evaluating treatment outcomes, designing intervention plans, and monitoring improvements in neck-related functionality.

SECONDARY OUTCOMES:
Range of Motion Measured by Goniometer | First day, after first week, after three weeks, after one month
  A goniometer is a standard instrument used to measure the range of motion (ROM) of the neck joints. It consists of arms and a protractor that allows clinicians to precisely quantify the angles achieved during various neck movements. During assessment, the patient is guided through specific motions like flexion, extension, rotation, and lateral bending, while the goniometer's arms are aligned with the corresponding body landmarks. The resulting measurements provide objective data about the neck's flexibility and mobility, aiding healthcare professionals in diagnosing musculoskeletal conditions, planning treatment strategies, and tracking progress over time.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa H Temel, M.D., Principal Investigator — Uskudar State Hospital

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be shared upon reasonable request by the principal investigator upon reasonable request.
Supporting Information: Study Protocol
Time Frame: 1 day
Access Criteria: The individual participant data will be shared upon reasonable request by the principal investigator upon reasonable request.